CLINICAL TRIAL: NCT03721783
Title: Infant and Child European Cryoablation Project ICECaP
Status: Recruiting | Type: Observational
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18BB37
Record Dates: First submitted 2018-10-10; First posted 2018-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Therapy; Soft Tissue Lesion; Cryoablation; Pediatric
Keywords: cryoablation; pediatric; registry
MeSH Terms: interventions — Cryosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children with soft tissue lesions: All children who undergo cryoablation therapy for benign soft tissue lesions
  Interventions: Procedure: Cryoablation

INTERVENTIONS:
Procedure: Cryoablation — Image guided cryoablation therapy of soft tissue lesions

SUMMARY:
A registry to audit the current range of applications, technical success rate, safety profile, complication rate and efficacy of cryoablation procedures being performed in children.

DETAILED DESCRIPTION:
Cryoablation involves image-guided insertion of single-use specialised needles or probes through the skin into a soft tissue or bone lesion. A mechanised unit is connected to the probe(s) and generates cyclical freezing and thawing of the tissues at the probe tip(s) via exchange of highly pressurised gases through the probe lumen(s), utilising the Joules-Thomson effect. Extreme freezing and thawing of the lesion causes permanent tissue destruction through both mechanical disruption of tissue membranes and a secondary immune response effect.

Cryoablation is one of several minimally invasive ablative techniques used to reduce the size of or to eradicate soft tissue and bone lesions. Ablative techniques are now an accepted standard of care for many benign and malignant lesions in adult practice. Cryoablation is widely used in the management of renal cell carcinoma, with medium-term outcomes matching surgical resection.

The advantages of cryoablation over surgery, particularly in a paediatric population, are:

* Minimally invasive approach, therefore suitable for day case procedures and almost scarless
* Significantly faster recovery times compared to complex surgical debulking
* Minimal complication rates compared to surgery (less risk to nerves, blood vessels and critical solid organ)
* Affords excellent pain relief (has an independent role in chronic pain management)

To date the use of cryoablation in children remains novel and under reported.

The purpose of this registry is to audit the current range of applications, technical success rate, safety profile, complication rate and efficacy of cryoablation procedures in children. This registry would, as a minimum, clarify current practice and outcomes within individual centres, allowing teams to audit and benchmark their own procedures and aiming to align practice amongst individual hospitals. A registry would aim to generate a body of evidence to establish parameters for best practice and may highlight conditions that respond better or worse than others to this novel therapy. The audit may lead to a clinical trial for the treatment of one or more specific conditions but in the interim would provide evidence for the efficacy and safety of the procedure and will aim to protect against indiscriminate use of this treatment modality in children in the future.

Registry design: This is a prospective multi-centre, open, non-controlled repeat treatment registry and data collection in collaboration with individual hospitals in the UK and Europe.

The proposal is for a robust, multi-centre data collection system to support and establish the treatment pathway, safety parameters and outcomes of paediatric cryoablation. The number of procedures performed in each centre will be understandably small, given the specialist nature of this emerging modality and the small numbers of patients being offered this treatment. The registry aims to collect standardised data from all centres performing cryoablation in children to allow robust audit of this procedure. Multiple data sets will be collected and entered into an anonymised web based host.

Upon completion of recruitment and follow up, the data will be subject to uni-variate and multi-variate analysis.

The registry is designed with the patient at the centre of the data collection and outcomes. Anonymised data will be analysed collectively but will ultimately be owned and retained by individual trusts. Details of the full data set proposed are detailed in the attached study protocol.

ELIGIBILITY:
Inclusion Criteria:

* all children in whom a clinical decision is made to treat with percutaneous cryoablation, to include those in whom cryoablation was not technically or clinically possible at any stage.

Exclusion Criteria:

* none

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children in whom a clinical decision is made to treat with percutaneous cryoablation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence and severity of complications arising from cryoablation treatment | 2 years
  Documentation and severity scoring of any complications arising from a cryoablation procedure, using the Society of Interventional Radiology (SIR) standards of practice committee classification of complications by outcome scoring system. The range of the outcome scoring system is A-F, with A being the least severe (no therapy, no consequence), and F being the most severe (resulting death). [Omary et al. J Vasc Interv Radiol 2003; 14:S293-S295]

SECONDARY OUTCOMES:
Change in maximal diameter of lesion following treatment | 5 years
  In patients where this is applicable, measure change in maximal lesion diameter on ultrasound or MRI imaging, comparing baseline (pre-treatment) lesion diameter to (post treatment) lesion diameter at 2 years. Subsequent lesion measurements will be made annually up to 5 years (for patients included in follow up).
Change in symptomatology following treatment | 2 years
  Where applicable, measure change in symptomatology post treatment, as assessed by PedsQL Pediatric Quality of Life Inventory UK questionnaire version 4.0. This is a scored questionnaire used for the assessment of physical functioning, emotional functioning, social functioning and school functioning. It is completed by both the child (child report) and the parent (parent report). Each questionnaire consists of 23 items graded 0-4 where 0 equates to no functional deficit and a maximum achievable score of 92 equates to the most severe functional deficit. Combined parent and child reports are collated to give a range of scores of 0-184 per assessment.
Procedure failure | 3 years
  This is a composite outcome defined as having the presence of any (or all) of the following: absence of consent, patient not fit for procedure, clinical complication, technical failure of equipment. This data will be collected over the 3 years of procedure recruitment into the registry.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Barnacle, BM, Principal Investigator — Great Ormond Street Hospital, London, UK
Locations (1):
- Great, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
This is planned as a multi centre registry, as there are other IR centres within the UK and Europe that wish to contribute paediatric data. This would be welcomed, to increase numbers and strengthen the outcome data

REFERENCES:
- [Result] Shaikh R, Alomari AI, Kerr CL, Miller P, Spencer SA. Cryoablation in fibro-adipose vascular anomaly (FAVA): a minimally invasive treatment option. Pediatr Radiol. 2016 Jul;46(8):1179-86. doi: 10.1007/s00247-016-3576-0. Epub 2016 Feb 22. PMID 26902298

DOCUMENTS (4):
  • Study Protocol: Appendix 1 security data protocol (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT03721783/Prot_001.pdf
  • Study Protocol: main document (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT03721783/Prot_004.pdf
  • Informed Consent Form: parent or guardian (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT03721783/ICF_005.pdf
  • Informed Consent Form: young person (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT03721783/ICF_006.pdf